CLINICAL TRIAL: NCT04657796
Title: Role of High Flow Nasal Oxygen as a Strategy for Weaning From Invasive Mechan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hamed Farag Qenawy Ahmed, Principal investigator, Assiut University
Other Study IDs: HFNCWEANINGMODE
Record Dates: First submitted 2020-10-04; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Failure With Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: High Flow Nasal Cannula — use of high flow nasal cannula as a weaning mode from invasive mechanical ventilation to deliver oxygen

SUMMARY:
evaluate the Efficacy of high flow nasal oxygen as a weaning strategy in mechanically ventilated patients with respiratory failure.

DETAILED DESCRIPTION:
Acute respiratory failure is a main cause of IMV and admission to intensive care unit (ICU){1}.

The day of extubation is a critical time during an intensive care unit (ICU) stay because in case of postextubation failure {2},which reach to 25 - 40% from extubated patient associated with VAP and barotrauma, mortality rate and hospital stay will increase , we use Adjuvant oxygen therapy to prevent these undesirable event like COT ,NIV and High-flow nasal cannula (HFNC) which can be used as an initial weaning strategy from IMVdue to its physiologic benefits [3-4].

HFNC devices supply between 30 and 60 L/min of a controlled mixture of actively warmed (32-37 °C) and humidified (up to 100% relative humidity) oxygen and air through modified nasal prongs. producing {5-6-7}:

1. moderate positive end-expiratory pressure (PEEP) .
2. HFNC might help prevent extubation failure through different

Mechanisms:

1. First, the controlled oxygen concentration may reduce transient hypoxemic episodes .
2. Second, the high flow washes the nasopharyngeal dead space, thus reducing CO2 re-breathing; this effect reduces respiratory rate and minute ventilation .
3. Third, the small amount of PEEP may reduce lung collapse . c)enabling better gas exchange and reduced work of breathing. d)in patients with chronic obstructive pulmonary disease (COPD), this level of PEEP may counterbalance auto PEEP, further reducing the work of breathing.

e) humidification may improve mucus drainage and reduce mucus retention, alleviating the associated atelectasis.

ELIGIBILITY:
Inclusion Criteria:

1- All adult patients who were admitted to our ICU requiring endotracheal intubation (ETI), were eligible for the study.

Exclusion Criteria:

1. Non-intubated patients or those with tracheostomy were excluded from the study.
2. those having neurological alteration unrelated to hypercapnoeic encephalopathy, cranio-facial deformity, upper airway obstruction, cardiogenic pulmonary edema, cardiogenic shock, acute myocardial infarction, pneumothorax, pulmonary neoplasm, pulmonary thromboembolism, gastrointestinal bleeding, and post-operative respiratory failure.
3. Patients less than 18 y.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient in respiratory ICU who mechanically intubated will be enrolled in study by using high flow nasal oxygen as a weaning strategy.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2020-12-05 (Estimated); Primary Completion 2022-10-05 (Estimated); Study Completion 2023-12-04 (Estimated)

PRIMARY OUTCOMES:
Is patient outcome in terms of survival or death at discharge. | through study completion average 7 days.
  evaluate the Efficacy of high flow nasal oxygen as a weaning strategy in mechanically ventilated patients with respiratory failure as regarding Hospitalization ,complications, oxygenation , reintubation rate, mortality rate.

SECONDARY OUTCOMES:
Duration of ICU stay through study completion average 7 days ,Adverse events. | through study completion average 7 days.
  evaluate efficacy of high flow nasal cannula on duration of hospital stay, complications rate.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Sl Sayed, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papazian L, Corley A, Hess D, Fraser JF, Frat JP, Guitton C, Jaber S, Maggiore SM, Nava S, Rello J, Ricard JD, Stephan F, Trisolini R, Azoulay E. Use of high-flow nasal cannula oxygenation in ICU adults: a narrative review. Intensive Care Med. 2016 Sep;42(9):1336-49. doi: 10.1007/s00134-016-4277-8. Epub 2016 Mar 11. PMID 26969671
- [Background] Helviz Y, Einav S. A Systematic Review of the High-flow Nasal Cannula for Adult Patients. Crit Care. 2018 Mar 20;22(1):71. doi: 10.1186/s13054-018-1990-4. PMID 29558988
- [Result] Drake MG. High-Flow Nasal Cannula Oxygen in Adults: An Evidence-based Assessment. Ann Am Thorac Soc. 2018 Feb;15(2):145-155. doi: 10.1513/AnnalsATS.201707-548FR. PMID 29144160